CLINICAL TRIAL: NCT07121556
Title: Randomized Double- Blind Study on the Treatment of Symptomatic Bilateral Knee Osteoarthritis: Intra-articular Injection of Autologous Microfragmented Adipose Tissue and Hyaluronic Acid vs Intra Articular Injection of Autologous Microfragmented Adipose Tissue. Double-Blind Randomized Controlled Clinical Trial
Brief Title: Treatment of Symptomatic Bilateral Knee Osteoarthritis: Intra-articular Injection of Autologous Microfragmented Adipose Tissue and Hyaluronic Acid vs Intra Articular Injection of Autologous Microfragmented Adipose Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HYALOFAT
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis Knees Both
Keywords: Osteoarthritis; Knees; HA; Micro-fragmented autologous adipose tissue; Hyaluronic acid; Intra-articular injection; Randomized double-blind study
MeSH Terms: conditions — Osteoarthritis | interventions — long-chain-alcohol O-fatty-acyltransferase

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled double-blind parallel-arm study with 1:1 allocation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient will not be aware of the side where hyaluronic acid will also be injected in addition to the microfragmented adipose tissue Clinical evaluations will be performed by medical personnel other than those who have performed the surgical and infiltrative procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFAT + HA left knee - MFAT + placebo right knee (Experimental): The left knee will be treated with an injection of high-molecular-weight hyaluronic acid (4 cc) and microfragmented autologous adipose tissue (6 cc), harvested from the abdominal site.The right knee will be treated with microfragmented autologous adipose tissue (6 cc), also harvested from the abdominal site by liposuction and microfragmentation, combined with an injection of 4 cc of saline (NaCl 0.9%)
  Interventions: Device: MFAT + HA left knee - MFAT + placebo right knee
- MFAT + HA right knee - MFAT + placebo left knee (Active Comparator): The right knee will be treated with an injection of high-molecular-weight hyaluronic acid (4 cc) and microfragmented autologous adipose tissue (6 cc), harvested from the abdominal site.The left knee will be treated with microfragmented autologous adipose tissue (6 cc), also harvested from the abdominal site by liposuction and microfragmentation, combined with an injection of 4 cc of saline (NaCl 0.9%)
  Interventions: Biological: MFAT + HA right knee - MFAT + placebo left knee

INTERVENTIONS:
Device: MFAT + HA left knee - MFAT + placebo right knee — The left knee will be treated with an injection of high-molecular-weight hyaluronic acid (4 cc) and microfragmented autologous adipose tissue (6 cc), harvested from the abdominal site.The right knee will be treated with microfragmented autologous adipose tissue (6 cc), also harvested from the abdominal site by liposuction and microfragmentation, combined with an injection of 4 cc of saline (NaCl 0.9%)
  Arms: MFAT + HA left knee - MFAT + placebo right knee
Biological: MFAT + HA right knee - MFAT + placebo left knee — The right knee will be treated with an injection of high-molecular-weight hyaluronic acid (4 cc) and microfragmented autologous adipose tissue (6 cc), harvested from the abdominal site.The left knee will be treated with microfragmented autologous adipose tissue (6 cc), also harvested from the abdominal site by liposuction and microfragmentation, combined with an injection of 4 cc of saline (NaCl 0.9%)
  Arms: MFAT + HA right knee - MFAT + placebo left knee

SUMMARY:
The HYALOFAT study is a randomized controlled double-blind trial with parallel treatment arms and 1:1 allocation.

By means of a double-blind randomized controlled trial in patients with symptomatic bilateral OA of the knees, the clinical outcomes of autologous microfragmented adipose tissue injection associated with hyaluronic acid in one knee vs autologous microfragmented adipose tissue injection in the contralateral knee will be evaluated and compared. Each patient will then serve as his or her own control and not be informed of the knee assigned to the treatment group. In addition, it will be the aim of the study to evaluate the safety of the combined treatment by documenting any adverse events.

DETAILED DESCRIPTION:
100 patients with symptomatic bilateral knee OA will be included in a randomized controlled double-blind study in which the clinical outcomes of treating OA with microfragmented autologous adipose tissue associated with high-molecular-weight hyaluronic acid versus treatment with microfragmented autologous adipose tissue will be evaluated and compared. One knee will be treated with an injection of high-molecular-weight hyaluronic acid (4 cc) and microfragmented autologous adipose tissue (6 cc), harvested from the abdominal site. The contralateral knee will be treated with microfragmented autologous adipose tissue (6 cc), also harvested from the abdominal site by liposuction and microfragmentation, combining an injection of 4 cc of saline (NaCl 0.9%) to make the volume of product injected into both knees equal. During screening, the eligibility of potentially enrollable subjects will be assessed.Once they are deemed eligible, the baseline visit will be performed, which will take place in the divisional or research clinic.

This will include: - the presentation of the study, the collection of informed consents and the administration and collection of subjective and objective evaluation questionnaires by medical staff. Patients will be clinically evaluated at 0-2-6-12 and 24 months follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 and 75;
2. Radiographic evidence of bilateral OA of the knees graded between 2 and 4 on the Kellgren-Lawrence scale;
3. Pain equal to or greater than 4 on the Numeric Rating Scale (NRS) for both knees;
4. Failure, defined as persistence of symptoms after at least 6 months of conservative treatment (pharmacological, physiotherapy, or infiltration treatment);
5. Ability and willingness to undergo the study procedures and comply with the instructions given by the study team; 6. No history of

4. Failure, defined as persistent symptoms, after at least 6 months of conservative treatment (pharmacological, physiotherapy, or infiltration treatment); 5. Ability and consent of patients to actively participate in the rehabilitation and follow-up protocol; 6. Signature of informed consent

Exclusion Criteria:

1. Patients incapable of understanding and willing;
2. Diagnosis of active neoplasia;
3. Diagnosis of rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis resulting from another inflammatory disease; human immunodeficiency virus (HIV) infection, active viral hepatitis; chondrocalcinosis;
4. Patients with uncontrolled diabetes mellitus;
5. Patients with uncontrolled thyroid metabolic disorders;
6. Patients who abuse alcohol, drugs, or medications;
7. Patients with lower limb misalignment greater than 5°;
8. Body Mass Index > 35 kg/m2;
9. Pregnancy or breastfeeding, or plans to become pregnant during the study period .
10. Patients with a history of trauma or intra-articular infiltration of therapeutic substances in the 6 months prior to screening.
11. Patients who have undergone knee surgery in the 12 months prior to screening.
12. Patients with insufficient abdominal adipose tissue, as assessed by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 months
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 2,6,24 months
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome
IKDC-Subjective Score | baseline, 2,6,12,24 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function.
IKDC-Objective Score (Objective International Knee Documentation Committee) | baseline, 2,6,12,24 months
  The objective assessment scale has seven parameters related to knee function. The presence of effusion and degree of knee movement are assessed, with the worst value of one of these parameters determining the final IKDC grade. There are four grades (A, B, C, D) which identify a knee assessed as normal, near normal, abnormal, and severely abnormal, respectively.
Patient Acceptable Symptom State (PASS) | baseline, 2,6,12,24 months
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
EuroQol Visual Analogue Scale (EQ-VAS) | baseline, 2,6,12,24 months
  EQ-VAS is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
Functional Numerical Rating Scale (NRS -functional) | baseline, 2,6,12,24 months
  It is a one-dimensional quantitative numerical scale for assessing functional impairment on a scale of 11 points; the scale requires the patient to select the number that best describes their state of functional disability, from 0 to 10. The higher the value indicated, the higher the degree of disability.
Numerical Rating Scale (NRS - pain) | baseline, 2,6,12,24 months
  It is a one-dimensional quantitative 11-point pain assessment scale; the scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that precise moment: 0 means no pain and 10 indicates the worst possible pain.
Objective parameters- Range of Motion | baseline, 2,6,12,24 months
  Evaluation of the Range of Motion for comparative analysis.
Objective parameters - Circumferences | baseline, 2,6,12,24 months
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis
Patient expectations regarding treatment | baseline
  The patient must indicate at baseline what clinical benefits they expect from the treatment according to the question: "What benefits do you expect to obtain from the treatment you will undergo?" The patient can choose from one of the following options: "complete recovery," "much better," "very much better," "a little better," or "no change."
Opinion on the treatment | 6,12,24 months
  The patient must indicate their level of satisfaction with the treatment received. The patient can choose from one of the following options: "much better," "a little better," "no change," "a little worse," and "much worse."
Effectiveness of the blinding procedure | baseline
  The patient is asked the following question: "In which knee do you think the treatment (autologous adipose tissue + hyaluronic acid) was performed?"
Safety of the procedure | baseline, 2,6,12,24 months
  The characteristics and incidence of any adverse events will be documented.
Medical history | baseline
  Recording of data relating to the duration and onset of symptoms, previous operations,level of activity, and cause of injury

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Martino, MD, Principal Investigator — Istituto Ortopedico Rizzoli - II Clinica Ortopedica e Traumatologica
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Holzbauer M, Priglinger E, Kolle ST, Prantl L, Stadler C, Winkler PW, Gotterbarm T, Duscher D. Intra-Articular Application of Autologous, Fat-Derived Orthobiologics in the Treatment of Knee Osteoarthritis: A Systematic Review. Cells. 2024 Apr 25;13(9):750. doi: 10.3390/cells13090750. PMID 38727286
- [Background] Bianchi F, Maioli M, Leonardi E, Olivi E, Pasquinelli G, Valente S, Mendez AJ, Ricordi C, Raffaini M, Tremolada C, Ventura C. A new nonenzymatic method and device to obtain a fat tissue derivative highly enriched in pericyte-like elements by mild mechanical forces from human lipoaspirates. Cell Transplant. 2013;22(11):2063-77. doi: 10.3727/096368912X657855. Epub 2012 Oct 8. PMID 23051701
- [Background] Tremolada C, Palmieri G, Ricordi C. Adipocyte transplantation and stem cells: plastic surgery meets regenerative medicine. Cell Transplant. 2010;19(10):1217-23. doi: 10.3727/096368910X507187. Epub 2010 May 4. PMID 20444320
- [Background] Perdisa F, Gostynska N, Roffi A, Filardo G, Marcacci M, Kon E. Adipose-Derived Mesenchymal Stem Cells for the Treatment of Articular Cartilage: A Systematic Review on Preclinical and Clinical Evidence. Stem Cells Int. 2015;2015:597652. doi: 10.1155/2015/597652. Epub 2015 Jul 9. PMID 26240572
- [Background] Van Pham P, Hong-Thien Bui K, Quoc Ngo D, Tan Khuat L, Kim Phan N. Transplantation of Nonexpanded Adipose Stromal Vascular Fraction and Platelet-Rich Plasma for Articular Cartilage Injury Treatment in Mice Model. J Med Eng. 2013;2013:832396. doi: 10.1155/2013/832396. Epub 2013 Jan 16. PMID 27006923
- [Background] Jurgens WJ, Kroeze RJ, Zandieh-Doulabi B, van Dijk A, Renders GA, Smit TH, van Milligen FJ, Ritt MJ, Helder MN. One-step surgical procedure for the treatment of osteochondral defects with adipose-derived stem cells in a caprine knee defect: a pilot study. Biores Open Access. 2013 Aug;2(4):315-25. doi: 10.1089/biores.2013.0024. PMID 23914338
- [Background] Filardo G, Tschon M, Perdisa F, Brogini S, Cavallo C, Desando G, Giavaresi G, Grigolo B, Martini L, Nicoli Aldini N, Roffi A, Fini M, Kon E. Micro-fragmentation is a valid alternative to cell expansion and enzymatic digestion of adipose tissue for the treatment of knee osteoarthritis: a comparative preclinical study. Knee Surg Sports Traumatol Arthrosc. 2022 Mar;30(3):773-781. doi: 10.1007/s00167-020-06373-y. Epub 2021 Jan 19. PMID 33464397
- [Background] Perucca Orfei C, Boffa A, Sourugeon Y, Laver L, Magalon J, Sanchez M, Tischer T, Filardo G, de Girolamo L. Cell-based therapies have disease-modifying effects on osteoarthritis in animal models. A systematic review by the ESSKA Orthobiologic Initiative. Part 1: adipose tissue-derived cell-based injectable therapies. Knee Surg Sports Traumatol Arthrosc. 2023 Feb;31(2):641-655. doi: 10.1007/s00167-022-07063-7. Epub 2022 Sep 14. PMID 36104484
- [Background] Vezzani B, Shaw I, Lesme H, Yong L, Khan N, Tremolada C, Peault B. Higher Pericyte Content and Secretory Activity of Microfragmented Human Adipose Tissue Compared to Enzymatically Derived Stromal Vascular Fraction. Stem Cells Transl Med. 2018 Dec;7(12):876-886. doi: 10.1002/sctm.18-0051. Epub 2018 Sep 26. PMID 30255987
- [Background] Desando G, Bartolotti I, Martini L, Giavaresi G, Nicoli Aldini N, Fini M, Roffi A, Perdisa F, Filardo G, Kon E, Grigolo B. Regenerative Features of Adipose Tissue for Osteoarthritis Treatment in a Rabbit Model: Enzymatic Digestion Versus Mechanical Disruption. Int J Mol Sci. 2019 May 29;20(11):2636. doi: 10.3390/ijms20112636. PMID 31146351
- [Background] Pak J. Regeneration of human bones in hip osteonecrosis and human cartilage in knee osteoarthritis with autologous adipose-tissue-derived stem cells: a case series. J Med Case Rep. 2011 Jul 7;5:296. doi: 10.1186/1752-1947-5-296. PMID 21736710
- [Background] Zaffagnini S, Andriolo L, Boffa A, Poggi A, Cenacchi A, Busacca M, Kon E, Filardo G, Di Martino A. Microfragmented Adipose Tissue Versus Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis: A Prospective Randomized Controlled Trial at 2-Year Follow-up. Am J Sports Med. 2022 Sep;50(11):2881-2892. doi: 10.1177/03635465221115821. Epub 2022 Aug 19. PMID 35984721
- [Background] Veronesi F, Andriolo L, Salerno M, Boffa A, Giavaresi G, Filardo G. Adipose Tissue-Derived Minimally Manipulated Products versus Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis: A Systematic Review of Clinical Evidence and Meta-Analysis. J Clin Med. 2023 Dec 22;13(1):67. doi: 10.3390/jcm13010067. PMID 38202074
- [Background] Qiao X, Yan L, Feng Y, Li X, Zhang K, Lv Z, Xu C, Zhao S, Liu F, Yang X, Tian Z. Efficacy and safety of corticosteroids, hyaluronic acid, and PRP and combination therapy for knee osteoarthritis: a systematic review and network meta-analysis. BMC Musculoskelet Disord. 2023 Nov 30;24(1):926. doi: 10.1186/s12891-023-06925-6. PMID 38037038
- [Background] Howlader MAA, Almigdad A, Urmi JF, Ibrahim H. Efficacy and Safety of Hyaluronic Acid and Platelet-Rich Plasma Combination Therapy Versus Platelet-Rich Plasma Alone in Treating Knee Osteoarthritis: A Systematic Review. Cureus. 2023 Oct 18;15(10):e47256. doi: 10.7759/cureus.47256. eCollection 2023 Oct. PMID 38022237
- [Background] Corradetti B, Taraballi F, Martinez JO, Minardi S, Basu N, Bauza G, Evangelopoulos M, Powell S, Corbo C, Tasciotti E. Hyaluronic acid coatings as a simple and efficient approach to improve MSC homing toward the site of inflammation. Sci Rep. 2017 Aug 11;7(1):7991. doi: 10.1038/s41598-017-08687-3. PMID 28801676
- [Background] Li L, Duan X, Fan Z, Chen L, Xing F, Xu Z, Chen Q, Xiang Z. Mesenchymal Stem Cells in Combination with Hyaluronic Acid for Articular Cartilage Defects. Sci Rep. 2018 Jul 2;8(1):9900. doi: 10.1038/s41598-018-27737-y. PMID 29967404
- [Background] Auw Yang KG, Raijmakers NJ, van Arkel ER, Caron JJ, Rijk PC, Willems WJ, Zijl JA, Verbout AJ, Dhert WJ, Saris DB. Autologous interleukin-1 receptor antagonist improves function and symptoms in osteoarthritis when compared to placebo in a prospective randomized controlled trial. Osteoarthritis Cartilage. 2008 Apr;16(4):498-505. doi: 10.1016/j.joca.2007.07.008. Epub 2007 Sep 6. PMID 17825587
- [Background] Bellamy N, Hochberg M, Tubach F, Martin-Mola E, Awada H, Bombardier C, Hajjaj-Hassouni N, Logeart I, Matucci-Cerinic M, van de Laar M, van der Heijde D, Dougados M. Development of multinational definitions of minimal clinically important improvement and patient acceptable symptomatic state in osteoarthritis. Arthritis Care Res (Hoboken). 2015 Jul;67(7):972-80. doi: 10.1002/acr.22538. PMID 25581339